CLINICAL TRIAL: NCT07099716
Title: Physiological Data Recording Over 24 Hours Using the Continual Optical Hilo Blood Pressure Monitor and an Ambulatory Blood Pressure Monitor: a Single-center, Prospective Clinical Study.
Brief Title: OBPM_HARMONY: Physiological Data Recording Over 24 Hours Using the Continual Optical Hilo Blood Pressure Monitor and an Ambulatory Blood Pressure Monitor
Acronym: OBPM_HARMONY
Status: Not yet recruiting | Type: Observational
Sponsor: Aktiia SA (Industry)
Responsible Party: Sponsor
Other Study IDs: OBPM_HARMONY
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
Keywords: HARMONY; Hypertension; CHUV
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Harmony study cohort: 24-hour Blood Pressure and Heart Rate monitoring with Hilo Band and Ambulatory Blood Pressure Monitor, in parallel of a 24-hour hydrostatic pressure monitoring for the same period
  Interventions: Device: Wearing Hilo band, Ambulatory Blood Pressure Monitor, and Hydrostatic Pressure monitor

INTERVENTIONS:
Device: Wearing Hilo band, Ambulatory Blood Pressure Monitor, and Hydrostatic Pressure monitor — During study Visit 1, participants are equipped with tthree devices- the Device Under Test (Hilo band), the reference device (Ambulatory Blood Pressure Monitor), worn on the opposite arm, and a Hydrostatic pressure monitor on the chest. Subjects are instructed to wear the three devices for the next 24 hours to collect blood pressure (BP) and heart rate (HR) data as well as hydrostatic pressure measurements. After Visit 1, subjects return home with the devices in place. Visit 2 takes place at least 24.5 hours later, when participants return to the site to hand back the equipment.

SUMMARY:
The OBPM_HARMONY study will enroll a minimum of 300 participants at the CHUV site in Lausanne, Switzerland. Each participant will complete two study visits at CHUV, scheduled at least 24.5 hours apart. Between these visits, participants will be asked to wear both the Hilo band, an Ambulatory Blood Pressure Monitor (ABPM) as well as a hydrostatic pressure system continuously for a 24-hour period.

DETAILED DESCRIPTION:
The OBPM_HARMONY study will enroll a minimum of N= 300 participants. Each participant will complete two visits at the CHUV site in Lausanne, Switzerland: Visit 1 (~40 minutes) and Visit 2 (~15 minutes), spaced at least 24.5 hours apart. During Visit 1, participants are equipped with three devices- the Device Under Test (Hilo band), the reference device (Ambulatory Blood Pressure Monitor), worn on the opposite arm, and a hydrostatic pressure system on the chest. Subjects are instructed to wear the three devices for the next 24 hours to collect blood pressure (BP) and heart rate (HR) data, as well as hydrostatic pressure measurements. After Visit 1, subjects return home with the devices in place. Visit 2 takes place at least 24.5 hours later, when participants return to the site to hand back the equipment and complete a feedback survey regarding their experience using the Hilo band and the ABPM reference.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 21 to 85yo
* Subjects fluent in written and spoken French, capable of discernment
* Subjects agreeing to attend the two study visits and follow study procedures
* Subjects residing within 100 km of the CHUV site
* Subjects that have signed the informed consent form.

Exclusion Criteria

* Damaged/injured skin at the right wrist
* Subjects with tachycardia (heart rate at rest > 120bpm)
* Subjects with atrial fibrillation
* Subjects with diabetes
* Subjects with marked renal dysfunctions
* Subjects with untreated hyper-/hypothyroidism
* Subjects with pheochromocytoma
* Subjects with Raynaud's disease
* Subjects with an arteriovenous fistula
* Subjects with implanted electrical devices, such as cardiac pacemakers or defibrillators
* Subjects with premature ventricular beats
* Subjects with peripheral arterial disease
* Subjects undergoing intravascular therapy or arterio-venous shunt
* Subjects who have received a mastectomy
* Women in known pregnancy or women with pre-eclampsia
* Subjects of unsound mind
* Subjects with upper arm circumference < 22cm or > 42cm
* Subjects with wrist circumference <14cm or > 23cm
* A lateral difference in systolic blood pressure >15 mmHg or diastolic blood pressure >10 mmHg between arms.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients attending the Nephrology and Hypertension Department at CHUV in Lausanne, Switzerland, for a consultation who, as part of their routine clinical care, require an Ambulatory Blood Pressure Monitor placement and meet the study's eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Raw 24-hour data collection using the continual Hilo monitor alongside the Ambulatory Blood Pressure Monitor across minimum 300 study subjects. | 24 hours

SECONDARY OUTCOMES:
Evaluation of survey results on comfort, usability, and ease of use for both devices | 24 hours

IPD SHARING:
Plan to Share IPD: Undecided